CLINICAL TRIAL: NCT01788267
Title: Evaluation of the Bone Microarchitecture in a Young Cystic Fibrosis Patients Using High-Resolution Peripheral Quantitative Computed Tomography
Brief Title: Bone Microarchitecture in Young Cystic Fibrosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011.678
Record Dates: First submitted 2013-02-05; First posted 2013-02-11 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2015-05

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; High-Resolution peripheral Quantitative Computed Tomography; Bone Mass Density
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy volunteers (Experimental): Volunteers realize a HR-pQCT scanner
  Interventions: Other: scan examination HR-pQCT
- Cystic Fibrosis patient (Experimental): Patients realize a HR-pQCT scanner
  Interventions: Other: scan examination HR-pQCT

INTERVENTIONS:
Other: scan examination HR-pQCT

SUMMARY:
Patients with cystic fibrosis are at risk of developing low bone mineral density (BMD) potentially leading to pathological fractures at adult age. Recent data from our center and others have suggested that low BMD could be observed very early in life. However, quantitative bone abnormalities found out by Dual X-ray absorptiometry (DXA) need to be confronted to qualitative evaluation of bone microarchitecture (surrogate of bone strength).

High-Resolution peripheral quantitative computed tomography (HR-pQCT) is a recent technology with very high spatial resolution. Images obtained with this technic are considered as virtual bone biopsies. It enables an accurate bones' cortical and trabecular surfaces exploration in a three-dimensional manner, and therefore provides informations on bone microarchitecture as well as bone density.

The aim of this study is to evaluate bone microarchitecture of paediatric patients matched to sex-age-pubertal status-healthy volunteers. In the meantime, biological markers will be collected and DXA (Dual-energy x-ray absorptiometry) will be performed in order to explore potential correlations HR-pQCT parameters.

ELIGIBILITY:
Inclusion Criteria:

* Cystic Fibrosis patient of both sex
* Pubertal patient
* Age ≥10 years and ≤18 years on the date of informed consent
* FEV1(forced expiratory volume at one second ) ≥ 60% of predicted normal for age, gender and height
* Patient on a clinical stable period

Exclusion Criteria:

* Unable to maintain arm and/or leg immobile for 3 minutes
* History of solid organ transplantation
* Participation in the same time to a clinical trial
* Acute pulmonary exacerbation at the time of evaluation

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Total Tibial Bone Mass Density measured by High-Resolution peripheral Quantitative Computed Tomography | at the inclusion visit J0

SECONDARY OUTCOMES:
total radial bone mass density | at the inclusion visit J0
Trabecular bone micro-architecture at tibia and radial sites | at the inclusion visit J0
Biological markers : 1) bone markers : parathyroid hormone (PTH), Calcifediol (25(OH)D3), osteocalcin, Endocrinal markers : IGF-1 (insulin like growth factor ), IGFBP-3, leptin, adiponectin, visfatin, resistin | at the inclusion visit J0

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme-Mère-Enfant, Bron, France

REFERENCES:
- [Result] Braun C, Bacchetta J, Braillon P, Chapurlat R, Drai J, Reix P. Children and adolescents with cystic fibrosis display moderate bone microarchitecture abnormalities: data from high-resolution peripheral quantitative computed tomography. Osteoporos Int. 2017 Nov;28(11):3179-3188. doi: 10.1007/s00198-017-4179-9. Epub 2017 Aug 9. PMID 28795206